CLINICAL TRIAL: NCT02638987
Title: EMG Activity, Muscle Tone, Elasticity and Stiffness of the Upper Trapezius Before, During and After Dry Needling
Brief Title: EMG Activity Before, During and After Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015/0740
Record Dates: First submitted 2015-12-09; First posted 2015-12-23 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Neck Pain
Keywords: Dry needling; office workers; myofascial pain; electromyography
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry needling (Experimental): After the second computer task, a single dry needling session will be performed with the subject lying on the non painful side. After palpation of a taut band and detection of MTrP 2 in the upper trapezius muscle, a trained physiotherapist will penetrate the needle into the MTrP and will move the needle up and down in multiple directions. When local twitch responses are elicited, this will be repeated until the local twitch responses are extinct.
  Interventions: Procedure: Dry needling
- Rest (No Intervention): After the first computer task, participants will rest in sidelying position for 10 minutes.

INTERVENTIONS:
Procedure: Dry needling — Dry needling (DN) is a myofascial treatment technique, in which a thin, solid filiform needle is inserted directly into the MTrP. During dry needling, local twitch responses (LTR) can be elicited. These are involuntary contractions of muscle fibers, leading to muscle relaxation, an increase in blood flow,recovery of the muscle metabolism and thus a reduction of pain and stiffness.
  Arms: Dry needling

SUMMARY:
An experimental study will be conducted to evaluate the effect of a single dry needling session on surface EMG activity (primary outcome measure), muscle tone, elasticity, stiffness and pain (secondary outcome measures) of the upper trapezius, in female office workers with trapezius myalgia.

DETAILED DESCRIPTION:
Neck-shoulder pain is a frequent problem in office workers . These complaints are often related to myofascial problems of neck and shoulder muscles in which the upper trapezius is frequently involved. Trapezius myalgia (TM) is characterized by pain, palpable stiffness and tenderness of the upper part of the trapezius muscle. Several studies show that myofascial trigger points (MTrP) have an important role in the development and maintenance of myofascial pain.

Trigger points are defined as hyperirritable nodules in a contracture of skeletal muscle fibers.

The pathophysiology of MTrPs is still unclear but several hypothesis exist. The most plausible explanation is that, due to sustained postures or repetitive low-level tasks, a sustained irritation of motor end plates with an excessive release of acetylcholine arises. This may lead to a persistent sarcomere contraction, leading to an impaired blood circulation, a reduced oxygenation and energy depletion, sensitizing nociceptors and causing pain.

Dry needling (DN) is a myofascial treatment technique, in which a thin, solid filiform needle is inserted directly into the MTrP. During dry needling, local twitch responses (LTR) can be elicited. These are involuntary contractions of muscle fibers, leading to muscle relaxation, an increase in blood flow, recovery of the muscle metabolism and thus a reduction of pain and stiffness.

In this experimental study, 25 female office workers with trapezius myalgia are recruited from several work places with predominantly computer based tasks. These subjects have to perform at least 20 hours a week of computer work and this since at least one year. Subjects are included based on online questionnaires, a clinical examination of neck an shoulder and the presence of MTRP 2 in the upper trapezius. All participants will receive information and have to sign an informed consent form.

Participants will be subjected to baseline assessment which involves measuring resting surface EMG activity, muscle tone, stiffness, elasticity and pain. Then, subjects have to perform a computer task during 20 minutes while surface EMG activity will be measured every 5 minutes. After this computer task, all measurements will be repeated. After a resting period of 10 minutes, baseline measurements are repeated, followed by a computer task of 20 minutes and repetition of the same assessment. After this computer task, a single dry needling session of MTrP 2 of the upper trapezius will be performed bilaterally. During this treatment, surface EMG activity will be measured to captivate the EMG activity during local twitch responses.

This is followed by repeating the same measurements 1 and 10 minutes after dry needling.

ELIGIBILITY:
Inclusion Criteria:

* Performing office work since at least one year
* Performing computer based tasks for at least 20 hours a week
* NRS > or equal to 3/10
* Clinical diagnosis of trapezius myalgia
* Trapezius myalgia is work-related and thus aggravates during working day/week
* Presence of MTrP2 in the upper trapezius muscle (bilaterally)

Exclusion Criteria:

* Being in treatment during the study
* Traumatic injuries/surgery to neck and upper limb region
* Signs of cervical nerve root impingement
* Whiplash injury
* Cardiovascular, neurological, life threatening, systemic and metabolic diseases
* Diagnosis of fibromyalgia/chronic fatigue syndrome
* Shoulder pathology
* Coagulation disorders
* Pregnancy

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in surface resting EMG activity of the upper trapezius after dry needling as assessed by the EMG DTS device | Immediately after a typing task of 20 minutes, one minute after dry needling, 10 minutes after dry needling
  Device: Noraxon USA Desktop Direct Transmission System (DTS) for EMG
  Changes in resting EMG activity of the upper trapezius immediately after dry needling and 10 minutes after dry needling, compared to resting EMG activity after a typing task, will be measured by using surface electrodes placed bilaterally at the MTrP 2 location of the upper trapezius (halfway between C7 and the posterolateral edge of the acromion). The change in EMG activity after dry needling will be compared with the change in EMG activity after rest.
  Resting EMG activity will be expressed as a percentage of submaximal reference contractions of the upper trapezius (% reference contractions).

SECONDARY OUTCOMES:
Changes in surface resting EMG activity of the upper trapezius after rest as assessed by the EMG DTS device | Immediately after a typing task of 20 minutes, immediately after a resting pause of 10 minutes
  Device: Noraxon USA Desktop Direct Transmission System (DTS) for EMG
  Changes in resting EMG activity of the upper trapezius after a resting pause of 10 minutes (in sidelying position), compared to resting EMG activity after a typing task, will be measured by using surface electrodes placed bilaterally at the MTrP 2 location of the upper trapezius (halfway between C7 and the posterolateral edge of the acromion).
  Resting EMG activity will be expressed as a percentage of submaximal reference contractions of the upper trapezius (% reference contractions).
Changes in surface resting EMG activity of the upper trapezius during a fatiguing typing task of 20 minutes as assessed by the EMG DTS device | During the typing task, every five minutes EMG activity will be measured for 30 seconds
  Device: Noraxon USA Desktop Direct Transmission System (DTS) for EMG
  Changes in EMG activity of the upper trapezius during a typing task of 20 minutes, will be measured by using surface electrodes placed bilaterally at the MTrP 2 location of the upper trapezius (halfway between C7 and the posterolateral edge of the acromion).
  EMG activity during this typing task will be expressed as a percentage of submaximal reference contractions of the upper trapezius (% reference contractions).
Differences in active muscle tension of the upper trapezius (ratio between resting EMG activity in upright and lying position) between the (dominant) painful and heterolateral side, as assessed by the EMG DTS device | At baseline
  Device: Noraxon USA Desktop Direct Transmission System (DTS) for EMG
  Resting EMG activity will be measured by using surface electrodes placed bilaterally at the MTrP 2 location of the upper trapezius (halfway between C7 and the posterolateral edge of the acromion).
  Resting EMG activity will be measured during 30 seconds with the subject lying supine, then resting EMG activity will be measured during 30 seconds with the subject seated in upright position. A ratio of both measurements will be calculated to compare active muscle tension the (dominant) painful and heterolateral side.
  Resting EMG activity will be expressed as a percentage of submaximal reference contractions of the upper trapezius (% reference contractions).
Differences in muscle fatigue of the upper trapezius (ratio between resting EMG activity before and after a typing task of 20 minutes) between the (dominant) painful and heterolateral side, as assessed by the EMG DTS device | Before and after a typing task of 20 minutes
  Device: Noraxon USA Desktop Direct Transmission System (DTS) for EMG
  Resting EMG activity will be measured by using surface electrodes placed bilaterally at the MTrP 2 location of the upper trapezius (halfway between C7 and the posterolateral edge of the acromion).
  Resting EMG activity will be measured during 30 seconds before starting the typing task and immediately after the typing task of 20 minutes. A ratio of both measurements will be calculated to compare muscle fatigue between the (dominant) painful and heterolateral side.
  Resting EMG activity will be expressed as a percentage of submaximal reference contractions of the upper trapezius (% reference contractions).
Changes in muscle tone, stiffness and elasticity of the upper trapezius after dry needling as assessed by the MyotonPRO ® | Immediately after a typing task of 20 minutes, one minute after dry needling, 10 minutes after dry needling
  Device: MyotonPRO ®
  Changes in muscle tone, stiffness and elasticity of the upper trapezius immediately after dry needling and 10 minutes after dry needling, compared to muscle tone, stiffness and elasticity after a typing task, will be measured by using the MyotonPRO ® device. This is placed on the upper trapezius halfway between C7 and the posterolateral part of the acromion.
  Muscle tone is expressed in Hertz (Hz) and characterizes muscle tone in resting state Muscle elasticity is the logarithmic decrement of the natural oscillation of the muscle Muscle stiffness is expressed in N/m (Newton per meter) and represents the resistance of the muscle to contraction.
Changes in muscle tone, stiffness and elasticity of the upper trapezius after rest as assessed by the MyotonPRO ® | Immediately after a typing task of 20 minutes, immediately after 10 minutes of rest
  Device: MyotonPRO ®
  Changes in muscle tone, stiffness and elasticity of the upper trapezius immediately after dry needling and 10 minutes after dry needling, compared to muscle tone, stiffness and elasticity will be measured by using the MyotonPRO ® device, which is placed on the upper trapezius halfway between C7 and the posterolateral part of the acromion
  Muscle tone is expressed in Hertz (Hz) and characterizes muscle tone in resting state Muscle elasticity is the logarithmic decrement of the natural oscillation of the muscle Muscle stiffness is expressed in N/m (Newton per meter) and represents the resistance of the muscle to contraction.
Changes in muscle tone, stiffness and elasticity of the upper trapezius after a typing task, compared to baseline, as assessed by the MyotonPRO ® | Before and immediately after a typing task of 20 minutes
  Device: MyotonPRO ®
  Changes in muscle tone, stiffness and elasticity of the upper trapezius after a typing task of 20 minutes, compared to baseline will be measured by using the MyotonPRO ® device, which is placed on the upper trapezius halfway between C7 and the posterolateral part of the acromion
  Muscle tone is expressed in Hertz (Hz) and characterizes muscle tone in resting state Muscle elasticity is the logarithmic decrement of the natural oscillation of the muscle Muscle stiffness is expressed in N/m (Newton per meter) and represents the resistance of the muscle to contraction.
Differences in muscle tone, stiffness and elasticity of the upper trapezius between the (dominant) painful and heterolateral side, as assessed by the MyotonPRO ® | At baseline
  Device: MyotonPRO ®
  Differences in muscle tone, stiffness and elasticity of the upper trapezius between the (dominant) painful and heterolateral side will be measured by using the MyotonPRO ®, which is placed on the upper trapezius halfway between C7 and the posterolateral part of the acromion
  Muscle tone is expressed in Hertz (Hz) and characterizes muscle tone in resting state Muscle elasticity is the logarithmic decrement of the natural oscillation of the muscle Muscle stiffness is expressed in N/m (Newton per meter) and represents the resistance of the muscle to contraction.
Changes in pain score after dry needling as assessed by the numeric rating scale | Immediately after a typing task of 20 minutes, one minute after dry needling, 10 minutes after dry needling
  Subjects will have to report their actual pain complaints on a numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain) after a typing task, one minute after dry needling and 10 minutes after dry needling.
Changes in pain score after rest as assessed by the numeric rating scale | Immediately after a typing task of 20 minutes, immediately after 10 minutes of rest
  Subjects will have to report their actual pain complaints on a numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain) after a typing task of 20 minutes and after a resting pause of 10 minutes.
Changes in pain score after a typing task of 20 minutes as assessed by the numeric rating scale | Immediately before and after a typing task of 20 minutes
  Subjects will have to report their actual pain complaints on a numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain) before and after a typing task of 20 minutes.
Differences in pain score at baseline between the (dominant) painful side and heterolateral side | At baseline
  Subjects will have to report their actual pain complaints on a numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain) for the (dominant) painful and heterolateral side.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, PhD, Principal Investigator — University Ghent